CLINICAL TRIAL: NCT00806884
Title: Do Physiotherapy Joint and Muscle Movement (Musculoskeletal) Techniques Improve Posture, Pain, Sputum Clearance, Lung Function or Quality of Life During Admission for a Respiratory Exacerbation in Adults With Cystic Fibrosis?
Brief Title: Do Physiotherapy Techniques Improve Posture During Admission for a Chest Infection in Adults With Cystic Fibrosis?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Professor ME Hodson, Royal Brompton & Harefield NHS Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 08/H0708/25; 2008CF003B
Record Dates: First submitted 2008-12-10; First posted 2008-12-11 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2008-12

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Musculoskeletal Physiotherapy; Manual therapy; Posture; Pain
MeSH Terms: conditions — Cystic Fibrosis; Pain | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Arm1 (Other): Normal optimal medical and physiotherapy treatment
  Interventions: Other: Control group measurements
- Treatment Arm 2 (Experimental): Physiotherapy musculoskeletal interventions in addition to normal optimal medical and physiotherapy care
  Interventions: Other: Physiotherapy Musculoskeletal Treatment

INTERVENTIONS:
Other: Physiotherapy Musculoskeletal Treatment — Other: Physiotherapy Musculoskeletal Treatment Specific, gentle oscillatory mobilisations to the rib cage and thoracic spine of the subjects to improve joint alignment and mobility, and to reduce pain. Treatment of specific muscle dysfunction or tight muscle groups to further optimise muscle length and biomechanical relationships in the area , leading to improved efficiency of recruitment and improved power output. Postural education and awareness discussions to improve the subject's own joint alignment and ability in a functional manner. A short programme to reinforce the progress during the treatment sessions may be given.
  Other Names: manual therapy; Manual techniques; physiotherapy joint mobilisations; physical therapy joint mobilisations
  Arms: Treatment Arm 2
Other: Control group measurements — None other than control group measurements
  Arms: Control Arm1

SUMMARY:
Hypothesis: The addition of a series of musculoskeletal techniques to normal optimal care for the treatment of a respiratory exacerbation in inpatient adults with cystic fibrosis, will lead to further improvements in pain, posture, sputum clearance, lung function and quality of life.

DETAILED DESCRIPTION:
Experimental design

A prospective, single blind, randomised control trial.

Methods

50 subjects will be recruited by the admitting physiotherapists from the inpatient wards at Royal Brompton Hospital. Using stratified computer randomisation, the subjects will be allocated to either the control (no treatment group) or the treatment group. The randomisation will be carried out by an independent member of the Department of Cystic Fibrosis and the outcome measures recorded by an observer blind to the randomisation.

Method:

* Two key investigators will be involved in the study to perform the treatment intervention as outlined in the paragraphs below
* The subjects' records will be reviewed by the key investigators to ensure they meet the inclusion criteria
* Prospective subjects will be given written and verbal information about the project and be given 24 hours to consider entry to the study
* Subjects will give written consent to participate in the project. The top copy will be included in the patient's medical record and a copy placed in the patient's study file
* A letter will be written to the subject's General Practitioner outlining the purpose of the study and inviting him/her to make contact to discuss the study in more detail if there are any queries or concerns
* The subjects will be withdrawn if there is a clinical deterioration negating the inclusion criteria or they are discharged for further home intravenous antibiotic treatment
* Three independent observers (the senior & junior physiotherapists usually working with this patient group) will be trained to ensure good intra & inter-relater reliability in the recording of the measurements

Intervention for the treatment group:

The treatment group will receive the interventions on top of their usual chest physiotherapy and medical care. A treatment series of gentle joint and muscle movements (musculoskeletal interventions) will be undertaken by a physiotherapist, on alternate days for the duration of admission. The physiotherapy musculoskeletal assessment and intervention may last up to 45 minutes on alternate weekdays and may include one or a combination of the following techniques which are documented in populations with postural changes, thoracic stiffness, discomfort and/or pain:

* Specific, gentle oscillatory mobilisations to the rib cage and thoracic spine of the subjects to improve joint alignment and mobility, and to reduce pain. These techniques should optimise chest wall mechanics, improve the length-tension relationships of the muscles and normalise movement to dysfunctional areas (Maitland, Banks et al. 2001;Mulligan 2005)
* Treatment of specific muscle dysfunction or tight muscle groups to further optimise muscle length and biomechanical relationships in the area (Massery 2005), leading to improved efficiency of recruitment and improved power output (Travell & Simons 1983)
* Postural education and awareness discussions to improve the subject's own joint alignment and ability in a functional manner. A short programme to reinforce the progress during the treatment sessions consisting of no more than three specific stretching or strengthening exercises may be given.

Control Group:

The control group will receive their usual medical and physiotherapy management but no placebo intervention.

Data Collection:

The outcome measures will be undertaken by one of three independent observers to pre-agreed protocols, before the first intervention session, and before intervention sessions on day five, day ten and day of discharge. The questionnaires CF-38 and the Hospital Anxiety and Depression Scale will be completed on initiation and completion of the study.

Sample size calculation: The number of patients needed for this study was based on testing of posture before and after musculoskeletal intervention in the outpatient adult cystic fibrosis randomised controlled trial ("Do physiotherapy musculoskeletal techniques improve forced expiratory volume in one second (FEV1) in adults with cystic fibrosis?"; Ethics reference number: 06/Q0404/81). To test for a three point change in thoracic index at the 5% significance level, using a square-root of within-mean standard of error of three would require at least 50 patients to achieve 90% power.

Analysis

Statistical advice was given by Mr Michael Roughton, Statistician, Royal Brompton Hospital and Imperial College London. The data will be analysed using an appropriate test e.g. t-tests or Mann-Whitney tests.

The intra & inter-rater reliability and repeatability of the measurements, by the independent observers, will be determined using Bland Atman plots to ensure they lie within clinically acceptable limits of agreement.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cystic fibrosis (genotype or sweat sodium >70 millimoles per litre or sweat chloride of >60 millimoles per litre)
* 16 years of age or over
* Inpatient admission for respiratory exacerbation as defined by the Cystic Fibrosis Trust (Cystic Fibrosis Trust Antibiotic Group 2002)
* Inpatients able to stand for the measurement period without cardiovascular or respiratory compromise.

Exclusion Criteria:

* Current severe haemoptysis
* Low bone density (Z score < -3)(World Health Organisation Study Group 1994)
* Rib fractures
* Pregnancy
* Inability to give consent for treatment/ measurement
* Planned initiation or continuation of treatment in the home environment
* Current participation in another study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-06; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Thoracic index as measured by the flexicurve (Boyle, Bradley et al. 2008). | Day 0 of admission, Days 5,10 & prior to discharge

SECONDARY OUTCOMES:
Lung function: forced expiratory volume in one second (FEV1), forced vital capacity (FVC) | Days 0,5,10 & pre discharge
Pain assessment using a 10-centimetre visual analogue scale | Days 0,5,10 & pre discharge
Sputum weight | Days 0,5,10
Ease of sputum clearance using a 10-centimetre visual analogue scale | Days 0,5,10 & pre discharge
Quality of life - CF-38 questionnaire (Ethics reference number: 98-167) | Days 0 & pre discharge
Hospital Anxiety and Depression Scale (Zigmond & Snaith 1983) | Days 0 & pre discharge

CONTACTS AND LOCATIONS:
Overall Officials: Professor ME Hodson, Principal Investigator — Imperial College London
Locations (1):
- Royal Brompton Hospital, London, London, United Kingdom